CLINICAL TRIAL: NCT00245362
Title: A Phase II Trial of CG 8020 and CG 2505 in Patients With Nonresectable or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-0011
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-10

CONDITIONS: Metastatic Pancreatic Cancer; Nonresectable Pancreatic Cancer
Keywords: cancer vaccine; pancreatic cancer; metastatic pancreatic cancer; unresectable pancreatic cancer; immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Biological: CG 8020 and CG 2505

SUMMARY:
To evaluate the safety and effectiveness of CG8020 and CG2505.

DETAILED DESCRIPTION:
To evaluate clinical and laboratory safety of CG 8020 and CG 2505 and to evaluate the efficacy of CG 8020 and CG 2505 as measured by clinical benefit response, progression-free survival, survival and CA 19-9 serum marker levels in chemotherapy naive or experienced patients with nonresectable or metastatic adenocarcinoma of the pancreas

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of nonresectable or metastatic pancreatic adenocarcinoma
* Chemotherapy naïve or chemotherapy experienced pancreatic cancer

Exclusion Criteria:

* Prior cancer vaccines or gene therapy
* History of clinically significant autoimmune disease (eg, systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis, glomerulonephritis, or vasculitis)
* History of another malignancy in the past five years, except adequately treated non-melanomatous skin cancer or superficial bladder cancer or carcinoma-in-situ of the cervix, unless approved by the Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Study Completion 2004-06

PRIMARY OUTCOMES:
Safety
Efficacy measured by clinical benefit response
Progression-free survivial
Overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - US Oncology, Dallas, Texas